CLINICAL TRIAL: NCT05054621
Title: A Single-blind, Randomized Study to Evaluate the Immunogenicity of Heterologous Prime-boost COVID-19 Vaccine Schedule
Brief Title: Immunogenicity of COVID-19 Vaccine on Heterologous Schedule
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Heterologous_AZ_Medigen
Record Dates: First submitted 2021-09-13; First posted 2021-09-23 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Covid-19; Vaccine; Immunogenicity; Reactogenicity; Healthy
MeSH Terms: conditions — COVID-19 | interventions — ChAdOx1 nCoV-19; MVC-COV1901 vaccine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heterologous group (Experimental): 1st dose AZD1222, 2nd dose MVC-COV1901
  Interventions: Biological: Heterologous prime-boost schedule with AZD1222 and MVC-COV1901
- Homologous group (control) (Active Comparator): 1st dose AZD1222, 2nd dose AZD1222
  Interventions: Biological: Homologous prime-boost schedule with two doses of AZD1222

INTERVENTIONS:
Biological: Heterologous prime-boost schedule with AZD1222 and MVC-COV1901 — Participants will be divided into two subgroups according to the intervals, 28-42 days and 56-70 days, between the prime and booster doses.
  Arms: Heterologous group
Biological: Homologous prime-boost schedule with two doses of AZD1222 — Participants will be divided into two subgroups according to the intervals, 28-42 days and 56-70 days, between the prime and booster doses.
  Arms: Homologous group (control)

SUMMARY:
This is a prospective, single blinded randomized homologous/heterologous prime-boost vaccine clinical study, designed to assess the immunogenicity of heterologous prime-boost immunization with AZD1222 and MVC-COV1901 in adults.

Participants will be healthy adults at the age of 20-70 years who have had their first dose of COVID-19 vaccine, AZD1222. All eligible participants of 2 prime-boost interval strata (28 to 42, 56 to 70 days) will be 1:1 randomly assigned to receive a single dose of either:

* Homologous group: Intramuscular injection the same vaccine as their prime dose AZD1222
* Heterologous group: Medigen COVID-19 vaccine MVC-COV1901. The treatment phase of this study will be conducted in a single-blind fashion such that the subject will not know the identity of the subjects' study treatment assignment. After receiving the treatment, the participants will remain on study for 168 days following the boost vaccination.

For the study primary objective, immunogenicity will be assessed during the duration of the study, including serologic neutralizing antibody titer against SARS-CoV-2, serological quantification of binding antibody to SARS-CoV-2 antigen, SARS-CoV-2 antigen specific B cell and T cell frequencies and cytokine levels.

And Safety will be assessed during the duration of the study as follows:

* Solicited adverse events (AEs; local and systemic) will be assessed for 7 days following each vaccination (Day 0 through Day 7 for the boost vaccination).
* Unsolicited AEs will be recorded for 28 days following the boost vaccination.
* Serious adverse events (SAEs) will be recorded from signing of the informed consent form through Day 168.
* Adverse events of special interest (AESIs) will be recorded from the boost vaccination through Day 168.

This study is going to be conducted in a single medical center in Taiwan. An appropriate number of participants will be screened to achieve approximately 44 evaluable participants for each group. Participants in each group will be divided into two subgroups according to the intervals, 28-42 days and 56-70 days, between the prime and booster doses.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give written informed consent for participation in the trial.
2. Male or Female, aged from 20 to 70 years
3. Has received one dose of the AZD1222 within 28-70 days before randomization. Evidence of this will be gathered from medical history and/or medical records including the COVID-19 vaccine registration yellow card.
4. Female participant must:

   1. Be either of non-childbearing potential, i.e. surgically sterilized (defined as having undergone hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy; tubal ligation alone is not considered sufficient) or one year post-menopausal;
   2. Or, if of childbearing potential, be abstinent or agree to use medically effective contraception on enrolment continuously until 90 days after boost immunization of study intervention.

   Acceptable forms include:

   i. Implanted hormonal methods of contraception or placement of an intrauterine device or intrauterine system ii. Established use of hormonal methods (injectable, pill, patch or ring) combined with barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository c. Have a negative pregnancy test.
5. In the Investigator's opinion, is able and willing to comply with all trial requirements.

Exclusion Criteria:

-

The participant may not enter the trial if ANY of the following apply:

1. Previous receipt of two or more COVID-19 vaccine doses
2. History of anaphylaxis, severe allergic disease or reactions likely to be exacerbated by any component of study vaccines (e.g. hypersensitivity to the active substance or any of the listed ingredients of any study vaccine). This includes latex and polyethylene glycol/macrogol (PEG)
3. Pregnancy, lactation or willingness/intention to become pregnant within 3 months post boost vaccine
4. Malignancy requiring receipt of immunosuppressive chemotherapy or radiotherapy for treatment of solid organ cancer/hematological malignancy within the 6 months prior to enrolment.
5. Bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following intramuscular injections or venipuncture.
6. Suspected or known current alcohol or drug dependency.
7. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.
8. Insufficient level of language to undertake all study requirements in opinion of the Investigators.
9. Known HIV antibody positive.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Immunogenicity: Neutralizing antibody against SARS-CoV-2 | Day 28 after booster dose
  To determine if the immune response to heterologous prime-boost immunization with ChAdOx1 nCOV-19 (AZD1222) and MVC-COV1901 is non-inferior to homologous prime-boost immunization with ChAdOx1 nCOV-19, in enrolled adult participants

SECONDARY OUTCOMES:
Immunogenicity：Anti-SARS-CoV-2 Spike antibody | base line (Day 0) and during the intervention at day 10, 28, 56 and 168 after booster dose of vaccine
  Further determination of Anti-SARS-CoV-2 Spike antibodies in all participants to heterologous/homologous prime-boost immunization of COVID-19 vaccines
Adverse events | through study completion, 6 months.
  To evaluate the safety of heterologous & homologous prime-boost immunization of COVID-19 vaccines
Immunogenicity: Anti-SARS-CoV-2 Nucleocapsid antibody | base line (Day 0) and during the intervention at day 10, 28, 56 and 168 after booster dose of vaccine
  Further determination of immunogenicity of Anti-SARS-CoV-2 Nucleocapsid in all participants to heterologous/homologous prime-boost immunization of COVID-19 vaccines.
Immunogenicity: T cell immunity | baseline (Day 0) and during the. intervention at day 10 and 28 after booster dose of vaccine
  Further determination of T cellular immune responses by ELISpot in all participants to heterologous/homologous prime-boost immunization of COVID-19 vaccines.

CONTACTS AND LOCATIONS:
Locations (1):
- ChangGungMH, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Chen CJ, Yang LY, Chang WY, Huang YC, Chiu CH, Shih SR, Huang CG, Huang KA. A randomized controlled trial of heterologous ChAdOx1 nCoV-19 and recombinant subunit vaccine MVC-COV1901 against COVID-19. Nat Commun. 2022 Sep 17;13(1):5466. doi: 10.1038/s41467-022-33146-7. PMID 36115850